CLINICAL TRIAL: NCT06008522
Title: Determining the Safety and Feasibility of Optical Coherence Tomography and Near Infrared Fluorescence: a Prospective Pilot Intervention Study
Brief Title: Safety and Feasibility of Immuno-OCT
Acronym: DETOUR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 11258
Record Dates: First submitted 2023-06-15; First posted 2023-08-23 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Colon Carcinoma; Barrett Esophagus; Gastrointestinal Dysplasia
Keywords: optical coherence tomography
MeSH Terms: conditions — Colonic Neoplasms; Barrett Esophagus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OCT with IV in colorectal polyps (Experimental): OCT and FME imaging of Barret and colorectal lesions during endoscopy.
  Interventions: Drug: Bevacizumab-800CW

INTERVENTIONS:
Drug: Bevacizumab-800CW — Imaging of fluorescently labeled Bevacizumab-800CW using OCT.
  Other Names: OCT imaging

SUMMARY:
To improve detection of premalignant lesions in the gastrointestinal tract (the rectum and the esophagus) there is a need for better endoscopic visualization and the ability for targeted biopsies. The University Medical Center Groningen (UMCG) developed a fluorescent tracer by labelling the VEGF-A-targeting humanized monoclonal antibody bevacizumab, currently used in anti-cancer therapy, with the fluorescent dye bevacizumab-800CW (IRDye800CW). In several phase I studies and phase II studies, either completed or currently running, in the UMCG, the use of VEGF-A-guided near-infrared (NIR) fluorescence molecular endoscopy (FME) in combination with high-definition white light endoscopy (HD-WLE) shows an improved detection rate of early premalignant lesions. In this study the safety and feasibility of a next generation imaging system will be tested. This system uses immune optical coherence tomography (immuno-OCT) and near infrared fluorescence (NIRF) with the targeted tracer (Bevacizumab-800CW) for improvement of the detection of dysplastic lesions in Barret's esophagus (BE) and colorectal polyp detection. The system provides more depth information and can eventually be used without the guidance of the regular endoscopy system.

ELIGIBILITY:
Inclusion Criteria:

* Indication for a therapeutic endoscopy procedure (EMR or ESD);
* Age ≥ 18;
* Written informed consent.

Exclusion Criteria:

* Patients younger than 18 years old;
* Submucosal and invasive esophageal adenocarcinoma (EAC) or colorectal carcinoma (CRC);
* Radiation therapy for esophageal or colorectal cancer;
* History of infusion reactions to Bevacizumab or other monoclonal antibodies;
* Chemotherapy, immunotherapy or surgery 28 days before administration of the tracer;
* Non-adjustable hypertension;
* Medical or psychiatric conditions that compromise the patient's ability to give informed consent;
* Pregnancy or breastfeeding; a negative pregnancy test must be available for women of childbearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Device-related Events (ADEs) and Serious Adverse Device-related Events (SADEs) using immuno-OCT | during procedure
  Any events related to the device.

SECONDARY OUTCOMES:
Validation of the immuno-OCT system: FME | During procedure
  Validation of the immuno-OCT endoscopy results compared to fluorescence seen in FME imaging results.
Validation of OCT system: Ex vivo fluorescence imaging | During procedure
  Validation of the immuno-OCT endoscopy results compared to the correlation of ex vivo fluorescent signals to histopathological analysis results.
validation of OCT system: ex vivo immuno-OCT imaging | During procedure
  Validation of the immuno-OCT endoscopy results compared to the correlation of in vivo and ex vivo immuno-OCT imaging to histopathological analysis results.
validation of OCT system: immunohistochemistry | Once, as soon as possible after procedure
  Validation of the in vivo immune-OCT endoscopy results by comparing it to histopathological analysis results.

CONTACTS AND LOCATIONS:
Overall Officials: W.B. Nagengast, MD, PhD, PharmD, Principal Investigator — University Medical Center Groningen

IPD SHARING:
Plan to Share IPD: No